CLINICAL TRIAL: NCT05425199
Title: Effects of Habituation Exercises Versus Proprioceptive Training on Dizziness, Vertigo, Balance and Quality of Life in Benign Paroxysmal Positional Vertigo
Brief Title: Habituation Exercises Versus Proprioceptive Training in Benign Paroxysmal Positional Vertigo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/22/0221 Nirmal Javed
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Benign Paroxysmal Positional Vertigo
Keywords: Habituation exercises; Proprioceptive training; Vertigo; Dizziness; Balance; benign paroxysmal positional vertigo
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Vertigo; Dizziness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- habituation exercises (Experimental): head and eye movements first slowly then rapidly, head and body movements e.g., picking object from the ground standing and rotation in standing
  Interventions: Other: Habituation exercises + vestibular treatment
- proprioceptive training (Experimental): Single leg stance (right side) + Single leg stance (left side) Lifting of right knee as high as comfortable and then alternative knee Tandem walking ,Toe walking ,Heel walking
  Interventions: Other: proprioceptive training + vestibular therapy
- Conventional vestibular therapy (Active Comparator): Epley's Manuever
  Interventions: Other: conventional vestibular treatment

INTERVENTIONS:
Other: Habituation exercises + vestibular treatment — Exercises will include Intensity: 10 repetitions of each set Frequency= 3 sessions per week for 6 weeks.
  Time= 30 minutes
  Arms: habituation exercises
Other: proprioceptive training + vestibular therapy — Exercise protocol will include Time= total session of 30 minutes . Each exercise will be hold for 30 seconds . Frequency= 3 session per week for 6 weeks Intensity= 10 repetitions and 3 sets
  Arms: proprioceptive training
Other: conventional vestibular treatment — Epley's Manuever. Frequency= It will be performed once in a week . Time= 10-15 minutes per session
  Arms: Conventional vestibular therapy

SUMMARY:
The aim of this research is to compare the effects of habituation exercises versus proprioceptive training on vertigo, balance, dizziness and quality of life in the individuals having benign paroxysmal positional vertigo. A randomized controlled trial that will include total 39 participants .The first group will receive habituation exercises for six weeks, three times per week for thirty minutes, along with conventional vestibular rehabilitation therapy. The second group will receive proprioceptive training for six weeks, three times per week for 30 minutes, along with vestibular rehabilitation therapy. The third group will only receive vestibular rehabilitation therapy. Data collected will be analyzed through SPSS 25.

DETAILED DESCRIPTION:
Benign paroxysmal positional vertigo is the most common presentation of peripheral vestibular disorder characterized by features like vertigo, nausea, vomiting, imbalance and increased risk of fall . Among all vestibular disorders, BPPV accounts for almost 20% and mostly affects the female gender as compared to the male gender. This type of disorder mainly involves the remoteness of otoliths in the semi-circular canal; most commonly the posterior canal is involved.

A comparative study on posterior canal BPPV including modified Epley procedure alone and Epley procedure combined with vestibular rehabilitation. This cross sectional study illustrated that the results of Epley maneuver only were as same as effectual as with VRT(vestibular Rehabilitation therapy) by reducing the symptoms of residual unsteadiness in that particular population. Among all vertiginous disorders BPPV is most common. Vestibular rehabilitation was conducted as therapeutic option and its effects on balance and quality of life were being assessed. Dizziness Handicap Inventory was being used as outcome measure scale.

The difference in signs of dizziness and quality of life in benign paroxysmal positional vertigo were investigated. Three groups were taken including one with BPPV, the second one with balance deficits (non-BPPV) and the last group involved healthy participants. The study concluded that the patients with BPPV had reduced HRQOL (health related Quality of life), tiredness and increased risk of fall. Dizziness associated with bed mobility is an indicator for the need of diagnoses and treatment thus, repositioning maneuvers had good impact on reducing the severity.

The effects of conventional vestibular rehabilitation recurrence rates on benign paroxysmal positional vertigo aimed to find the impacts on otolith dysfunction. Although repositioning movements were proved fruitful yet the recurrence rates were high in older population as compared to young. Vestibular therapy including habituation exercises decreases the risks of recurrence in benign paroxysmal positional vertigo.

As balance impairments are common in individuals with vertigo and dizziness. Proprioceptive training was proved more efficient than vestibular therapy in reducing the chances of fall in elder population. BBS (berg balance scale) and TUG (Time up and Go test) were conducted to assess balance and risk of fall in older people.

Systematic review of the previous literature on the efficacy of vestibular rehabilitation therapy in benign paroxysmal positional vertigo.12 studies were based on inclusion criteria and the effectiveness of vestibular rehabilitation only and in combination with repositioning maneuver and also in comparison with it. Habituation exercises were included in VR therapeutic intervention, Conclusion were in favor of vestibular therapy as it showed reduction in discomfort caused by the condition.

Efficacy of vestibular therapy protocol to determine its effects on quality of life and postural balance. Randomized controlled trial was performed on 20 individuals. Outcome measure scales like DHI (dizziness handicap inventory), VAS (vertigo visual analogue scale) were used and it was observed that with vestibular rehabilitation there were consequences like better quality of life and reduced signs of vertigo and dizziness were achieved.

According to previous study there was a lack of control group in previous evidence whereas this study will focus on control as well as interventional groups. In previous literature, both of these therapeutic options i.e., habituation exercises and proprioceptive training were used in combination but in this study the comparison will be done between two exercise protocols.

Consequences will be manipulated for balance, vertigo, dizziness and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Chronic vestibular disorder
* Diagnosed BPPV patients
* Normal vision
* Score of > 1 on VAS for vertigo
* Score of > 50 on DHI questionnaire
* Ability to follow the command

Exclusion Criteria:

* CNS involvement
* Orthopedic problem
* Unable to answer a simple verbal command
* Head injury or brain trauma
* Not medically diagnosed with any vestibular disorder

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-06-05 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Berg balance scale | 6th week
  Consists of 14 tasks and total score of 56.score of 0-20 indicates severe fall risk, 20-45 includes moderate risk of fall and 45-60 illustrates thr functional balances state.

SECONDARY OUTCOMES:
dynamic gait index | 6th week
  Assess the likelihood of falling in older adults.total score is of 24.score less than 19 is predictive of fall risks.
Dizziness handicap inventory | 6th week
  Measure of patients perception of dizziness.subscales included are functional, physical and emotional.
visual vertigo analogue scale | 6th week
  This scale rates the intensity of visual vertigo in nine challenging situations of visual motions and categorized as having no (0), Mild (0.1-40), moderate (40.01-70) or severe (70.01-100) symptoms.
Activities specific balance confidence scale | 6th week
  Assess the older individuals balance confidence in performing daily life activities. This scale comprises of a wide continuum of less and more challenging activities.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Aabroo, Principal Investigator — Riphah International University
Locations (1):
- psrd (pakistan Society for the rehabilitation of the disabled, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marsden J, Pavlou M, Dennett R, Gibbon A, Knight-Lozano R, Jeu L, Flavell C, Freeman J, Bamiou DE, Harris C, Hawton A, Goodwin E, Jones B, Creanor S. Vestibular rehabilitation in multiple sclerosis: study protocol for a randomised controlled trial and cost-effectiveness analysis comparing customised with booklet based vestibular rehabilitation for vestibulopathy and a 12 month observational cohort study of the symptom reduction and recurrence rate following treatment for benign paroxysmal positional vertigo. BMC Neurol. 2020 Nov 27;20(1):430. doi: 10.1186/s12883-020-01983-y. PMID 33243182
- [Background] Bressi F, Vella P, Casale M, Moffa A, Sabatino L, Lopez MA, Carinci F, Papalia R, Salvinelli F, Sterzi S. Vestibular rehabilitation in benign paroxysmal positional vertigo: Reality or fiction? Int J Immunopathol Pharmacol. 2017 Jun;30(2):113-122. doi: 10.1177/0394632017709917. Epub 2017 May 9. PMID 28485653
- [Background] Rodrigues DL, Ledesma ALL, de Oliveira CAP, Bahamad Junior F. Physical Therapy for Posterior and Horizontal Canal Benign Paroxysmal Positional Vertigo: Long-term Effect and Recurrence: A Systematic Review. Int Arch Otorhinolaryngol. 2018 Oct;22(4):455-459. doi: 10.1055/s-0037-1604345. Epub 2017 Aug 28. PMID 30357032
- [Background] Roller RA, Hall CD. A speed-based approach to vestibular rehabilitation for peripheral vestibular hypofunction: A retrospective chart review. J Vestib Res. 2018;28(3-4):349-357. doi: 10.3233/VES-180633. PMID 29689764
- [Background] Bayat A, Saki N. Effects of Vestibular Rehabilitation Interventions in the Elderly with Chronic Unilateral Vestibular Hypofunction. Iran J Otorhinolaryngol. 2017 Jul;29(93):183-188. PMID 28819615
- [Background] Colnaghi S, Rezzani C, Gnesi M, Manfrin M, Quaglieri S, Nuti D, Mandala M, Monti MC, Versino M. Validation of the Italian Version of the Dizziness Handicap Inventory, the Situational Vertigo Questionnaire, and the Activity-Specific Balance Confidence Scale for Peripheral and Central Vestibular Symptoms. Front Neurol. 2017 Oct 10;8:528. doi: 10.3389/fneur.2017.00528. eCollection 2017. PMID 29066999
- [Background] Tramontano M, Martino Cinnera A, Manzari L, Tozzi FF, Caltagirone C, Morone G, Pompa A, Grasso MG. Vestibular rehabilitation has positive effects on balance, fatigue and activities of daily living in highly disabled multiple sclerosis people: A preliminary randomized controlled trial. Restor Neurol Neurosci. 2018;36(6):709-718. doi: 10.3233/RNN-180850. PMID 30412513
- [Background] Heydari M, Ahadi M, Jalaei B, Maarefvand M, Talebi H. The Additional Effect of Vestibular Rehabilitation Therapy on Residual Dizziness After Successful Modified Epley Procedure for Posterior Canal Benign Paroxysmal Positional Vertigo. Am J Audiol. 2021 Sep 10;30(3):535-543. doi: 10.1044/2021_AJA-20-00171. Epub 2021 Jun 30. PMID 34191552
- [Background] Lindell E, Kollen L, Johansson M, Karlsson T, Ryden L, Falk Erhag H, Wetterberg H, Zettergren A, Skoog I, Finizia C. Benign paroxysmal positional vertigo, dizziness, and health-related quality of life among older adults in a population-based setting. Eur Arch Otorhinolaryngol. 2021 May;278(5):1637-1644. doi: 10.1007/s00405-020-06357-1. Epub 2020 Sep 19. PMID 32948896
- [Background] Traboulsi H, Teixido M. Qualitative analysis of the Dix-Hallpike maneuver in multi-canal BPPV using a biomechanical model: Introduction of an expanded Dix-Hallpike maneuver for enhanced diagnosis of multi-canal BPPV. World J Otorhinolaryngol Head Neck Surg. 2017 Jun 8;3(3):163-168. doi: 10.1016/j.wjorl.2017.01.005. eCollection 2017 Sep. PMID 29516062